CLINICAL TRIAL: NCT01403389
Title: Pilot Study of the Clinical Activity of Eculizumab for Prevention of Delayed Graft Function in Patients Undergoing Deceased Donor Kidney Transplantation
Brief Title: A Study of the Activity of Eculizumab for Prevention of Delayed Graft Function In Deceased Donor Kidney Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After interim analysis, the pilot study was terminated and modified to a larger multicenter study (NCT01919346) to better assess efficacy.
Sponsor: Schroppel, Bernd, M.D. (Individual)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSM 10-1600
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Delayed Function of Renal Transplant
Keywords: Kidney Transplant; Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function | interventions — eculizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eculizumab (Experimental)
  Interventions: Drug: Eculizumab
- 0.9% Sodium Chloride (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eculizumab — 1200 milligrams Eculizumab diluted in 0.9% NaCl to 5mg/mL for a total volume of 240 mL administered by IV infusion over 35 minutes in the operating room prior to organ reperfusion
  Other Names: Soliris
  Arms: Eculizumab
Drug: Placebo — 240 mL of 0.9% Sodium Chloride IV fluid given as placebo in the operating room prior to organ reperfusion
  Other Names: 0.9% Sodium Chloride
  Arms: 0.9% Sodium Chloride

SUMMARY:
The purpose of this study is to determine if Eculizumab is safe and effective in the prevention of delayed graft function following deceased donor kidney transplantation.

DETAILED DESCRIPTION:
Based on experimental data and supportive observations in humans associating complement gene upregulation with ischemic reperfusion injury, it is hypothesized that C5 cleavage is a key step in the pathogenesis of ischemic reperfusion injury following transplantation. It is further hypothesized that eculizumab, an antibody that blocks C5 cleavage in humans will be an effective prophylactic agent to prevent ischemic reperfusion injury in high risk recipients. To test this hypothesis, this study is a pilot prospective, randomized study to test the efficacy of eculizumab vs. placebo given once at the time of transplantation in preventing delayed graft function in first adult recipients of deceased donor kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Weight > 40 kg
* Male or Female
* Recipients of first deceased donor kidneys
* Able to provide written informed consent
* Transplant candidate as per site specific guidelines
* Dialysis dependent renal failure (initiated more than 2 months prior to transplant)
* Novartis Delayed Graft Function Score 3-8
* Extended criteria donor with brain death, or standard criteria donor with cold ischemic time < 24 hours

Exclusion Criteria:

* Planned to receive multi-organ transplant
* Kidneys from donors < 6 years of age
* Dual kidney transplant (from same donor, including en bloc)
* Living donor kidney
* Highly sensitized recipients (PRA > 50%)
* Previous transplant
* Participation in another investigational trial
* Recipient BMI > 40
* ABO incompatible
* DCD Donor
* Preemptive kidney transplant
* Recipients with DGF scores < 3 or > 8
* Women who are pregnant or breast feeding
* Women of child bearing potential who are unable or unwilling to use a medically acceptable form of contraception
* Patients infected with HIV, HCV or HBV
* Active bacterial or other infection which is clinically significant in the opinion of the investigator
* Patients with history of splenectomy
* Patients with history of meningococcal disease
* Patients with known or suspected hereditary complement deficiency
* Patients with history of cancer (other than non-melanoma skin cancers) within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2013-08-06 (Actual); Study Completion 2014-02-06 (Actual)

PRIMARY OUTCOMES:
Composite of Delayed Graft Function and Slow Graft Function | Up to 6 months
  Delayed Graft Function defined as follows:
  1. A need for at least one dialysis treatment during the first 7 days after transplantation (not including a single session for hyperkalemia or hypervolemia in the first 48 hours)
  2. A less than or equal to 50% reduction in serum creatinine in the first 24 hours post-transplantation
  3. A serum creatinine reduction ratio < 30% at 48 hours post-transplantation
  Slow Graft Function Defined as Follows:
  A functioning graft at Day 5 Post-transplantation with a serum creatinine > 3 mg/dL and no need for dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Schroppel, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Recanati/Miller Transplantation Institute, New York, New York, United States